CLINICAL TRIAL: NCT05338346
Title: A Phase I, Open-Label, Multi-Center, Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG-018 (ATR Inhibitor) Treatment in Patients With Advanced Solid Tumors and Hematological Malignancies
Brief Title: A Study of ATG-018 (ATR Inhibitor) Treatment in Patients With Advanced Solid Tumors and Hematological Malignancies
Acronym: ATRIUM
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy of study compound
Sponsor: Antengene Discovery Limited (Industry)
Responsible Party: Sponsor
Organization: Antengene Corporation (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-018-001
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Advanced Solid Tumors; Hematological Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-018 (Experimental): Dose Escalation Phase:
  For Solid Tumors Group: A maximum of 44 subjects with solid tumors will be enrolled during the Dose Escalation Phase.
  For Hematological Malignancies Group: Subjects with hematological malignancy will be enrolled.
  Dose Expansion Phase:
  The tumor types in Dose Expansion Phase may involve other tumor types based on the signals from the Dose Escalation Phase. Each tumor type is planned to enroll at least 12 subjects, and a further expansion (up to 40 subjects in each tumor type) may be triggered if 2 or more confirmed responses are observed in this cohort.
  Interventions: Drug: ATG-018

INTERVENTIONS:
Drug: ATG-018 — Dose Escalation Phase:
  For both dose escalation groups, subjects will receive a single dose of ATG-018 monotherapy on Cycle 1 Day 1 (C1D1) for single dose PK samples' collection. From the morning dose on Cycle 1 Day 2, twice daily dosing (except Dose Level 1: 5 mg QD) will be initiated. Subject(s) will receive intermittent dosing in a 3 days on/4 days off schedule in 21-day cycles until disease progression or unacceptable toxicity.
  Dose Expansion Phase :
  Dose Expansion Phase will begin at the defined MTD/RP2D for solid tumors and hematological malignancies groups, to further evaluate the safety, tolerability, and PDx profile of ATG-018. Subjects with solid tumors and hematological malignancies will be enrolled.

SUMMARY:
This is a Phase I, Open-Label, Multi-Center, Dose Finding Study to Investigate the Safety, Pharmacokinetics, and Preliminary Efficacy of ATG-018 (ATR inhibitor) Treatment in Patients with Advanced Solid Tumors and Hematological Malignancies .

DETAILED DESCRIPTION:
This is a Phase I, multi-center, open-label study of ATG-018 administered orally as monotherapy in patients with advanced solid tumors and hematological malignancies. The study design includes a Dose Escalation Phase and a Dose Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all the following inclusion criteria to be eligible to enroll in this study:

  1. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling, and analyses.
  2. Aged at least 18 years.
  3. After completion of Dose level 3, subjects will need to demonstrate a defect in one or more DDR genes such as: ATM (including ATM protein loss by IHC), ATRX, ARID1A, BARD1, BRCA1, BRCA2, BRIP1, CDK12, CHEK2, FANCA, FANCC, FANCD2, FANCE, FANCF, FANCM, MRE11A, MSH2, NBN, PALB2, RAD51, RAD51B, RAD51C, RAD51D, or other related genes at the discretion of the investigator in consultation with sponsor Medical Monitor; Or mutations in p53 pathway/MYC pathway.
  4. Subjects with solid tumor must meet the following criteria: histological or cytological confirmation of a solid tumor, and have progressed despite standard therapy(ies), or are intolerant to standard therapy(ies), or have a tumor for which no standard therapy(ies) exists. Locally recurrent disease must not be amenable to surgical resection or radiotherapy with curative intent (subjects who are considered suitable for surgical or ablative techniques following down-staging with study treatment are not eligible).
  5. Subjects with hematological malignancies must meet the following criteria: have pathologically confirmed de novo DLBCL or DLBCL transformed from previously diagnosed indolent lymphoma (eg, follicular lymphoma) or B-cell indolent Non-Hodgkin's Lymphoma (iNHL) with histological subtype limited to FL Grade 1, Grade 2, or Grade 3a, or Grade 3b, or splenic marginal zone lymphoma (MZL), or nodal MZL, or extranodal MZL based on criteria established by the World Health Organization (WHO) 2016 classification.
  6. Subjects with DLBCL must have received at least 2 previous systemic regimens for the treatment of their de novo or transformed DLBCL including at least 1 course of anthracycline-based chemotherapy (unless absolutely contraindicated due to cardiac dysfunction, in which case other active agents such as etoposide, bendamustine, or gemcitabine must have been given) combined with at least 1 course of anti-CD20 immunotherapy (eg, rituximab), unless contraindicated due to severe toxicity. Prior stem cell transplantation was allowed; induction, consolidation, stem cell collection, preparative regimen, and transplantation ± maintenance were considered a single line of therapy.
  7. Subjects with B-cell iNHL must have received at least one previous line of therapy including a CD20-targeted monoclonal antibody, and systemic therapy does not include local involved field radiotherapy for limited stage disease and/or H. Pylori eradication.

     Please note that all hematological malignancies must have documented clinical or radiographic evidence of progressive prior to dosing.
  8. Subjects must have measurable lesion defined as below:

     1. Subject with solid tumors must have at least 1 lesion, not previously irradiated, that can be accurately measured at pre dose as ≥10 mm in the longest diameter (except lymph nodes which must have short axis ≥15 mm) with CT or MRI and which is suitable for accurate repeated measurements.
     2. Subject with B-NHL must have measurable disease as defined by at least one bi-dimensionally measurable lesion that node >1.5 cm in longest diameter (LDi) or extranodal lesion >1 cm in LDi (per the Lugano 2014 Criteria).
  9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 with no deterioration over the previous 2 weeks, or prior to the first dose of study treatment (C1D1).
  10. Except for hearing loss, alopecia, and pigmentation, all toxicity caused by previous antitumor therapy has recovered to Grade 1 or less (according to the NCI-CTCAE version 5.0).
  11. Life expectancy >3 months.
  12. Men and women of childbearing potential must agree to use effective contraceptives from they sign the informed consent to 180 days after the last dose of study drug. Women of childbearing potential include premenopausal women and women within 2 years after menopause. Women of childbearing age must have a negative serum pregnancy test at screening.
  13. Male subjects (including those who have undergone vasectomy) must consent to the use of condoms during sex with women of childbearing potential and have no plans to impregnate the woman during the use of the study drug and within 180 days after the last dose of the study drug from the date of signing the ICF.
  14. Subjects should have the ability and willingness to comply with the study and follow up.

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria are not eligible to enroll in this study:

  1. Central nervous system (CNS) metastatic disease, leptomeningeal disease, or metastatic cord compression.
  2. Prior treatment with ATR inhibitor.
  3. Subjects with B-NHL in the condition as below:

     1. DLBCL with MALT lymphoma.
     2. Composite lymphoma (Hodgkin's lymphoma + NHL).
     3. Primary mediastinal (thymic) large B-cell lymphoma.
  4. Prior therapy with any other investigational product or anticancer systemic therapy including chemotherapy, immunotherapy, or other anticancer agents within 21 days (or within a period during which the investigational product or systemic anticancer treatment has not been cleared from the body, eg, a period of 5 'half-lives') of the first dose of study treatment, whichever is the most appropriate as judged by the investigator.
  5. Radiotherapy with a wide field of radiation within 28 days, or radiotherapy with a limited field of radiation for palliation within 14 days of the first dose of study treatment. Subject must have recovered from all radiation related toxicity, not requiring corticosteroids.
  6. Prior major surgery (excluding placement of vascular access) within 28 days of the first dose of study treatment or minor surgical procedures ≤7 days. No waiting is required following implantable port and catheter placement.
  7. Subjects receiving unstable or increasing doses of corticosteroids. For patients receiving corticosteroids for endocrine deficiencies or symptoms associated to their disease (excluding central nervous system disease), the dose must have been stabilized (or reducing) for at least 14 days before the first dose of study treatment.
  8. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension defined as a blood pressure (BP) ≥150/95 mmHg despite medical therapy, unstable or uncompensated respiratory and renal disease, active bleeding diseases, allogeneic stem cell transplantation, or any solid organ transplant.
  9. Have active or previous autoimmune diseases that are likely to recur (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, vasculitis, and psoriasis), or are at risk of such diseases.
  10. Poorly controlled of pleural effusion or pericardial effusion (with clinical symptoms, fluctuation of effusion or need for repeated drainage, oral diuretics, etc) at screening. Ascites that can be detected on physical examination, or clinical symptoms caused by ascites, or that require special treatment, such as repeated drainage, intraperitoneal drug infusion, etc, at screening (Subjects with a small amount of ascites that can only be detected by imaging examination can be considered for inclusion).
  11. Active infection including hepatitis B, and/or hepatitis C (HBV-DNA or HCV-RNA detected above lower limit of normal [LLN] by local laboratory, respectively).
  12. Known history of human immunodeficiency virus (HIV) infection.
  13. Active infection requiring parenteral antibiotics, antivirals, or antifungals within 14 days prior to C1D1; however, prophylactic use of these agents is acceptable (including parenteral).
  14. Autologous stem cell transplant < 6 months or CAR-T cell infusion < 6 months prior to C1D1.
  15. History of allogeneic stem cell transplant.
  16. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

      1. Unstable angina or acute myocardial infarction ≤3 months prior to C1D1.
      2. Clinically significant heart disease (eg, symptomatic congestive heart failure with New York Heart Association Grade 3 or above).
      3. Uncontrolled arrhythmia, or hypertension; history of labile hypertension or poor compliance with an antihypertensive regimen.
      4. Baseline left ventricular ejection fraction (LVEF) below institution's LLN or <50% if assessed by echocardiogram (ECHO), or baseline LVEF below institution's LLN if assessed by multiple gated acquisition scan (MUGA).
  17. Inadequate bone marrow reserve (within 14 days) or organ function as demonstrated by any of the following laboratory values:

      1. Absolute neutrophil count <1.5 × 109/L
      2. Platelet count <100 × 109/L
      3. Hemoglobin <90 g/L Please note that platelet transfusions within 7 days, red blood cell transfusions within 14 days, hematopoietic growth factors within 7 days (G-CSF or erythropoietin) are not permitted prior to obtaining these laboratory values.

      <!-- -->

      1. Alanine aminotransferase (ALT) >2.5 times the upper limit of normal (ULN)
      2. Aspartate aminotransferase (AST) >2.5 times ULN
      3. Total bilirubin >1.5 times ULN
      4. Creatinine >1.5 times ULN concurrent with creatinine clearance <50 mL/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN

      <!-- -->

      1. Serum albumin <30 g/L
      2. Coagulation: international normalized ratio (INR) >2.0, prothrombin time (PT) >1.5×ULN
  18. Subject inability or unwillingness to comply with requirement for oral drug administration or presence of a gastro-intestinal condition, eg, refractory nausea and vomiting, any acute or chronic gastrointestinal disease, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of ATG-018.
  19. History of hypersensitivity to any excipient of ATG-018 or these medicinal products or history of allergic reactions attributed to drugs with a similar chemical structure or class to ATG-018.
  20. Any chronic or uncontrolled dermatological condition that will be adversely impacted by the potential skin toxicity of the study treatment(s).
  21. Judgment by the investigator that the subject should not participate in the study if the subject is unlikely to comply with study procedures, restrictions, and requirements.
  22. Other primary malignancies developed within 2 years prior to the first administration of the study drug, except locally curable malignancies after radical treatment (such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast, etc).
  23. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
  24. Subjects was in receipt of any live attenuated vaccination within 30 days prior to the first dose of study treatment.
  25. History or current evidence of any condition or disease that could confound the results of the study or, in the opinion of investigator, is not in the best interest of the subject to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-01-08 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
AE/SAE | 12 months after the last subject enrolled
  Adverse Event/Serious Adverse Event
MTD | 12 months after the last subject enrolled
  Maximum Tolerated Dose
RP2D | 12 months after the last subject enrolled
  RP2D= Recommended Phase 2 Dose

SECONDARY OUTCOMES:
ORR | 12 months after the last subject enrolled
  Overall Response Rate
DOR | 12 months after the last subject enrolled
  Duration of Response

OTHER OUTCOMES:
PFS | 12 months after the last subject enrolled
  Progression Free Survival
OS | 12 months after the last subject enrolled
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Icon Cancer Centre South Brisbane, Brisbane
  - Chris O'Brien Lifehouse, Camperdown
  - Austin Health, Heidelberg
  - Alfred Health, Melbourne
  - Liverpool Hospital, Sydney